CLINICAL TRIAL: NCT06355011
Title: Total Elbow Replacement in England: Analysis of National Joint Registry and Hospital Episode Statistics Data
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: The National Joint Registry (Unknown); The Royal College of Surgeons of England (Other); John Charnley Trust (Unknown); University of Bristol (Other)
Responsible Party: Principal Investigator, Zaid Hamoodi, National Joint Registry research fellow and PhD Student, University of Manchester
Other Study IDs: 7016194
Record Dates: First submitted 2024-03-19; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Total Elbow Replacement
MeSH Terms: interventions — Arthroplasty, Replacement, Elbow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Total Elbow Replacement — Total elbow replacement is a procedure that involves replacing the elbow joint with an implanted device to alleviate pain and improve function.

SUMMARY:
The goal of this observational registry study is to provide detailed descriptions of the patients who are receiving primary total elbow replacement surgery in England. The main questions it aims to answer are:

* Who are receiving primary total elbow replacement surgery?
* Where and by whom is the total elbow replacement surgery is being performed?
* What the current surgical practices for total elbow replacement?

Pseudonymous data from the National Joint Registry NJR of all patients with total elbow replacement will be used.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 to 100 years old with a primary TER on the National Joint Registry (NJR) elbow dataset from the start of data collection on the 1st of April 2012 to the 31st of December 2022 will be included.

Exclusion Criteria:

* Patients are excluded if they did not consent for their data to be used for research purposes, if it is impossible to trace them after surgery, if their ID numbers are invalid, or if the surgery was not performed in England.
* Unconfirmed procedures and procedures with inconsistent operative patterns (i.e. a sequence of operations where the primary operation is not the first operation in the sequence or where there are multiple primary operations recorded for the same joint) will be excluded from the analyses.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a primary total elbow replacement in England on the National Joint Registry (NJR)
Sampling Method: Non-Probability Sample
Enrollment: 3891 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
The incidence of total elbow replacement (TER) in England | Yearly (1 year) incidence for a 10 year period
  The number and age-sex standardised rate of TER for different sexes, ethnicities, and socioeconomic backgrounds.

SECONDARY OUTCOMES:
Serious adverse events or re-admissions | 30 and 90 days after the index TER
  Serious adverse events will be defined as any severe medical complications leading to hospital admission, including pulmonary embolism, myocardial infarction, lower respiratory tract infection, acute kidney injury, urinary tract infection, cerebrovascular events, and all-cause death.
Duration of elective wait | Up to 10 years period
  The number of days between the decision for total elbow replacement and the actual day of surgery
Post-operative duration of stay | Up to 10 years period
  The number of days from the time of surgery until discharge from the hospital
Surgeon volume | 10 year (2012 to 2022)
  Number of TERs performed by a surgeon per year by surgeons in England
Hospital volume | 10 year (2012 to 2022)
  Number of TERs performed by a hospital per year by surgeons in England

OTHER OUTCOMES:
Patient characteristics (Age) | 10 year (2012 to 2022)
  Age in years
Body mass index | 10 year (2012 to 2022)
  BMI measured in in kg/m^2
Hand dominance | 10 year (2012 to 2022)
  Dominant non-dominant hand
American Society of Anaesthesiologists (ASA) grade | 10 year (2012 to 2022)
  Grades 1-5
Indication for total elbow replacement | 10 year (2012 to 2022)
  Categories: Acute trauma/inflammatory/ Trauma sequelae/Osteoarthritis/ Other
Socioeconomic status | 10 year (2012 to 2022)
  Categorical: Indices of multiple deprivation quintiles (2015 version)
Ethnicity | 10 year (2012 to 2022)
  Categorical: Asian, Asian British, or Asian Welsh /Black, Black British, Black Welsh, Caribbean or African/White/Mixed or Multiple ethnic groups/Other ethnic group
Co-morbidities | 10 year (2012 to 2022)
  Categorical: Acute MI /CHF / PVD/ Cerebrovascular Disease / Dementia/ COPD/ Rheumatoid Disease/ Peptic Ulcer/ Mild liver disease/ Diabetes/ Diabetes + Complications/ Hemiplegia or Paraplegia/ Renal disease/ Cancer/ Moderate/Severe liver disease/ Metastatic Cancer/ AIDS/ Depression/ Anxiety/ Osteoporosis
Charlson Comorbidity Index | 10 year (2012 to 2022)
  Original Charlson Comorbidity Index
Implant classification | 10 year (2012 to 2022)
  Categorical: Linked/ Unlinked
Fixation type | 10 year (2012 to 2022)
  Categorical: Cemented/ Uncemented
Implant type | 10 year (2012 to 2022)
  Categorical: Coonrad-Morrey/ Discovery/ Latitude (Legacy, EV, Mix)/ GSB III/ MUTARS/ Nexel/ IBP
If radial head replacement was used | 10 year (2012 to 2022)
  Categorical: Yes/No
Grade of primary surgeon | 10 year (2012 to 2022)
  Categorical: Consultant/Other
Funding | 10 year (2012 to 2022)
  Categorical: National Health Services (NHS) /Independent sector
Elective admission type | 10 year (2012 to 2022)
  Categorical: General admission/ Day case admission

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Epidemiology Versus Arthritis, Centre for Musculoskeletal Research, University of Manchester, Manchester Academic Health Science Centre, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The National Joint Registry (NJR) elbow data can be requested for research purposes through an application to the NJR research committee. Researchers do not have the rights to share the data directly

REFERENCES:
- [Derived] Hamoodi Z, Sayers A, Whitehouse MR, Rangan A, Kearsley-Fleet L, Sergeant JC, Watts AC. Total elbow replacement in England: a protocol for analysis of National Joint Registry and Hospital Episode Statistics data. J Orthop Surg Res. 2024 Aug 30;19(1):526. doi: 10.1186/s13018-024-04903-9. PMID 39215301